CLINICAL TRIAL: NCT03717012
Title: Study of Pulmonary Rehabilitation In Nintedanib Treated Patients With IPF: Improvements in Activity, Exercise Endurance Time, and QoL
Brief Title: Study of Pulmonary Rehabilitation in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated prematurely due to difficulties with recruitment because of the COVID-19 pandemic.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0324
Expanded Access: NCT03843892 (Approved for marketing)
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nintedanib treatment alone (Active Comparator)
  Interventions: Drug: Nintedanib
- Nintedanib with a pulmonary rehabilitation program (Experimental)
  Interventions: Drug: Nintedanib; Other: Pulmonary rehabilitation program

INTERVENTIONS:
Drug: Nintedanib — stable dose
Other: Pulmonary rehabilitation program — 12 weeks
  Arms: Nintedanib with a pulmonary rehabilitation program

SUMMARY:
The main objectives of this study are:

* Determine the difference in change from baseline in Six Minute Walk Distance (6MWD) when pulmonary rehabilitation (PR) is added to stable underlying nintedanib therapy in patients with idiopathic pulmonary fibrosis (IPF)
* Determine the difference in change in Quality of Life (QoL) when pulmonary rehabilitation (PR) is added to stable underlying nintedanib therapy in patients with idiopathic pulmonary fibrosis (IPF)
* Determine if there is an enduring effect in 6MWD, QoL and lung function from pulmonary rehabilitation (PR) when pulmonary rehabilitation (PR) is added to stable underlying nintedanib therapy in patients with idiopathic pulmonary fibrosis (IPF)

ELIGIBILITY:
Inclusion criteria:

* Patients being treated with a stable dose of nintedanib 150 mg BID for up to 30 months. Patients who have recently started nintedanib 150 mg BID and have started by the day of randomization must be on nintedanib 150 mg BID a minimum of 10 days by the first day of pulmonary rehabilitation.
* Age ≥ 40 years at screening
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient consent form
* Signed and dated written informed consent in accordance with ICH-GCP (International Council on Harmonization and Good Clinical Practice) and local legislation prior to admission to the trial
* Confirmed diagnosis of IPF according to 2011 American Thoracic Society (ATS)/ European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guidelines by lung biopsy or High Resolution Computed Tomography (HRCT)(based upon INPULSIS criteria, (if biopsy only or HRCT done > 24 months prior to screening, a new HRCT to be done after consent and prior to or up to 7 days after Visit 2 for quantitative lung fibrosis score (QLF) for disease characterization)
* Forced Vital Capacity (FVC) ≥ 45% of predicted by the NHANES equation or equivalent (after discussion with Clinical Monitor), historical within past 30 days can be used. Carbon monoxide Diffusion Capacity (DLCO) (corrected for hemoglobin [Hgb]) 30-79% of predicted
* FEV1/FVC greater than/equal to .7
* Physically capable of performing both a 6 minute walk test and work rate cycle ergometry (sub-study patients), must successfully complete the practice tests for the 6 minute walk test, per the instructions. Potential sub-study patients that require supplemental oxygen or cannot complete the incremental work rate cycle ergometry test will not participate in the sub-study, but will qualify for the main study.

Exclusion criteria:

* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned within 6 months after screening, e.g. hip replacement which could interfere with the ability to participate in pulmonary rehabilitation.
* Any documented active or suspected malignancy or history of malignancy within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous enrolment in this trial (except for rescreening)
* Currently enrolled in another interventional investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial
* Women who are pregnant, nursing, or who plan to become pregnant in the trial
* Previous participation in pulmonary rehabilitation program within 45 days prior to signing consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - Western Connecticut Medical Group, Danbury, Connecticut
  - Miami VA Healthcare System, Miami, Florida
  - Coastal Pulmonary & Crit Care, St. Petersburg, Florida
  - The LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - Pulmonary and Critical Care Associates of Baltimore, Towson, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - St. Vincent Physicians Sleep and Respiratory Center, Billings, Montana
  - Glacier View Research Institute, Kalispell, Montana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Pulmonix, LLC, Greensboro, North Carolina
  - Temple University Hospital, Oaks, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Metroplex Pul and Sleep Ctr, McKinney, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, open-label, prospective, Phase IV clinical trial of pulmonary rehabilitation during the first 12 weeks of a 24-week treatment period, compared with no pulmonary rehabilitation, in patients already taking nintedanib for idiopathic pulmonary fibrosis.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Nintedanib 150 mg: Subjects were required to be treated on a stable (up to 30 months) dose of nintedanib 150 milligram (mg) twice a day (BID) administered per prescribing instructions and to continue on this dose throughout the trial. Patients who recently started nintedanib 150 mg BID and have started by the day of randomization must be on nintedanib 150 mg BID a minimum of 10 days by the first day of pulmonary rehabilitation. Patients that have had an interruption in nintedanib treatment or a temporary dose reduction can be entered into the trial when they have returned to a dose of 150 mg BID and their condition is determined to be stable by the investigator and temporary dose reductions to treat adverse events is permitted during the trial.
- Nintedanib 150 mg + Pulmonary Rehabilitation: Subjects were required to be treated on a stable (up to 30 months) dose of nintedanib 150 milligram (mg) twice a day (BID) administered per prescribing instructions and to continue on this dose throughout the trial. Patients who recently started nintedanib 150 mg BID and have started by the day of randomization must be on nintedanib 150 mg BID a minimum of 10 days by the first day of pulmonary rehabilitation. Patients that have had an interruption in nintedanib treatment or a temporary dose reduction can be entered into the trial when they have returned to a dose of 150 mg BID and their condition is determined to be stable by the investigator and temporary dose reductions to treat adverse events is permitted during the trial.
  In addition patients received a standard pulmonary rehabilitation regimen two or three times weekly for 12 weeks. The pulmonary rehabilitation should follow the facility's standard regimen as long as the regimen meets basic standards.
Period: Overall Study
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Started | 9 | 10
Completed | 8 | 4
Not Completed | 1 | 6
Not completed — Due to trial termination | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lung transplant | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set (RS): This patient set includes all randomized patients, whether treated with pulmonary rehabilitation or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.5) | 70.9 (11.9) | 69.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
6 minute walk distance (6MWD) test [Mean (Standard Deviation); unit: meter] — 6 minute walk distance (6MWD) test at baseline. The last assessment before treatment period start (included) will be used as baseline. If the baseline value is missing and the screening value is available, then the baseline value will be defined as the screening value taken closest to baseline date.
  meter | 360 (159.03) | 322.33 (114.30) | 340.17 (134.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 6 Minute Walk Test (6MWD) at 12 Weeks
Description: Absolute change from baseline in the 6 minute walk distance (6MWD) test at 12 weeks. The last assessment before treatment period start (included) will be used as baseline. If the baseline value is missing and the screening value is available, then the baseline value will be defined as the screening value taken closest to baseline date.
Time Frame: Baseline (day 1) and week 12 (day 85).
Population: Randomized set (RS): This patient set includes all randomized patients, whether treated with pulmonary rehabilitation or not.
  Patients with no data available at week 12 were excluded.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
meter | -20.60 (31.24) | -14.10 (53.99)

2. Secondary Outcome: Change From Baseline in the 6 Minute Walk Test (6MWD) at 24 Weeks
Description: Absolute change from baseline in the 6 minute walk distance (6MWD) test at 24 weeks. The last assessment before treatment period start (included) will be used as baseline. If the baseline value is missing and the screening value is available, then the baseline value will be defined as the screening value taken closest to baseline date.
Time Frame: Baseline (day 1) and week 24 (day 169).
Population: Randomized set (RS): This patient set includes all randomized patients, whether treated with pulmonary rehabilitation or not.
  Patients with no data available at week 24 were excluded.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 5 | 3
meter | -38.34 (63.24) | 9.04 (10.82)

3. Secondary Outcome: Change From Baseline in the St George's Respiratory Questionnaire (SGRQ) Total Score at 12 and 24 Weeks
Description: Absolute change from baseline in the St George's Respiratory Questionnaire (SGRQ) total score at 12 and 24 weeks. The SGRQ is a widely used disease specific questionnaire evaluating health related quality of life. The SGRQ Total Score is measured using patient self-reported question on disease impact on symptoms, patient activity, and daily life. SGRQ scores are calculated using weights attached to each item of the questionnaire which provides an estimate of the distress associated with the symptoms or state described in each item. The total score for SGRQ ranges from 0 to 100, with higher scores indicating more limitations.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: Randomized set (RS): This patient set includes all randomized patients, whether treated with pulmonary rehabilitation or not.
  Patients with no data available at week 12 or week 24 were excluded from their respective analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Score on a scale.
  Change from baseline at week 12 | 5.60 (11.43) | -1.48 (9.03)
  Change from baseline at week 24: number analyzed (Participants) | 6 | 3
  Change from baseline at week 24 | 6.06 (13.38) | -6.54 (4.97)

4. Secondary Outcome: Absolute Change From Baseline in The King's Brief Interstitial Lung Disease (KBILD) Questionnaire Total Score at 12 and 24 Weeks
Description: Absolute change from baseline in The King's Brief Interstitial Lung Disease (KBILD) questionnaire total score at 12 and 24 weeks. The KBILD questionnaire is a disease specific questionnaire evaluating health related quality of life. The questionnaire consists of 15 items. Raw total scores were weighted with a Likert response scale to create the total score, total scores were transformed to a range of 0-100 ((actual score-lowest possible score/range)*100), with a score of 100 representing the best health status.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Score on a scale.
  Change from baseline at week 12 | -3.20 (3.21) | 1.28 (5.36)
  Change from baseline at week 24: number analyzed (Participants) | 6 | 3
  Change from baseline at week 24 | -4.42 (8.80) | -0.63 (4.87)

5. Secondary Outcome: Change From Baseline in the University of California, San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) Total Score at 12 and 24 Weeks
Description: Change from baseline in the University of California, San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) total score at 12 and 24 weeks. The UCSD-SOBQ is a 24-item questionnaire that assesses self-reported shortness of breath while performing a variety of activities of daily living, scores for each item range from 0 to 5, with higher scores indicating more limitations. Total score is calculated as the sum of all individual scores. Scores range from 0 to 120, with higher scores indicating more limitations.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Score on a scale.
  Change from baseline at week 12 | 13.29 (12.63) | 6.13 (18.71)
  Change from baseline at week 24: number analyzed (Participants) | 6 | 3
  Change from baseline at week 24 | 17.50 (14.54) | 0.00 (19.97)

6. Secondary Outcome: Absolute Change From Baseline of Forced Vital Capacity (FVC) at 12 and 24 Weeks
Description: Absolute change from baseline of forced vital capacity (FVC) at 12 and 24 weeks. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Milliliter (mL)
  Change from baseline at week 12 | -152.86 (261.90) | -87.50 (277.32)
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24 | 76.00 (356.13) | -86.67 (168.62)

7. Secondary Outcome: Absolute Change From Baseline of Forced Vital Capacity (FVC) % Predicted at 12 and 24 Weeks
Description: Absolute change from baseline of forced vital capacity (FVC) % predicted at 12 and 24 weeks. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. For predicted normal values, different sites may use different prediction formulas, based on the method used to measure diffusing capacity of the lung for carbon monoxide (DLco). In any case, the method used must be in compliance with the European Respiratory Society (ERS)/American Thoracic Society (ATS) guideline on DLco measurements, and the prediction formula appropriate for that method.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Percent predicted
  Change from baseline at week 12 | -3.84 (7.93) | -1.50 (7.42)
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24 | 3.63 (11.69) | -1.93 (4.44)

8. Secondary Outcome: Relative Change From Baseline of Forced Vital Capacity (FVC) at 12 and 24 Weeks
Description: Relative change (unitless) from baseline of forced vital capacity (FVC) at 12 and 24 weeks. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC is measured in milliliter (mL). Its relative change from baseline at 12 (24) weeks is calculated as: (FVC measured at 12 (24) weeks - FVC measured at baseline)/ FVC measured at baseline *100%.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Percent change
  Change from baseline at week 12 | -3.68 (9.35) | -2.60 (9.02)
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24 | 2.80 (10.12) | -2.16 (4.64)

9. Secondary Outcome: Relative Change From Baseline of Forced Vital Capacity (FVC) % Predicted at 12 and 24 Weeks
Description: Relative change (unitless) from baseline of forced vital capacity (FVC) % predicted at 12 and 24 weeks. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. For predicted normal values, different sites may use different prediction formulas, based on the method used to measure diffusing capacity of the lung for carbon monoxide (DLco). In any case, the method used must be in compliance with the European Respiratory Society (ERS)/American Thoracic Society (ATS) guideline on DLco measurements, and the prediction formula appropriate for that method. The relative change from baseline of FVC % predicted at 12 (24) weeks is calculated as: (FVC % Predicted measured at 12 (24) weeks - FVC % Predicted measured at baseline)/ FVC % Predicted measured at baseline *100%.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Percent change
  Change from baseline at week 12 | -3.68 (9.35) | -2.60 (9.02)
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24 | 2.80 (10.12) | -2.16 (4.64)

10. Secondary Outcome: Absolute Categorical Change of Forced Vital Capacity (FVC)% Predicted up to 12 and 24 Weeks (Decrease by >5%, Increase by >5%, and Change Within ≤5%)
Description: Absolute categorical change of forced vital capacity (FVC)% predicted up to 12 and 24 weeks, the following three categories were defined: decrease by >5%, increase by >5%, and change within ≤5%. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. For predicted normal values, different sites may use different prediction formulas, based on the method used to measure diffusing capacity of the lung for carbon monoxide (DLco). In any case, the method used must be in compliance with the European Respiratory Society (ERS)/American Thoracic Society(ATS) guideline on DLco measurements, and the prediction formula appropriate for that method.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Participants
  Change from baseline at week 12: Decrease by >5% | 4 | 2
  Change from baseline at week 12: Within 5% change | 2 | 5
  Change from baseline at week 12: Increase by >5% | 1 | 1
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24: Decrease by >5% | 1 | 1
  Change from baseline at week 24: Within 5% change | 2 | 2
  Change from baseline at week 24: Increase by >5% | 2 | 0

11. Secondary Outcome: Absolute Categorical Change of Forced Vital Capacity (FVC)% Predicted up to 12 and 24 Weeks (Decrease by >10%, Increase by >10%, and Change Within ≤10%)
Description: Absolute categorical change of forced vital capacity (FVC)% predicted up to 12 and 24 weeks, the following three categories were defined: decrease by >10%, increase by >10%, and change within ≤10%. Forced Vital Capacity (FVC) is the volume of air (measured in milliliter) which can be forcibly exhaled from the lungs after taking the deepest breath possible. For predicted normal values, different sites may use different prediction formulas, based on the method used to measure diffusing capacity of the lung for carbon monoxide (DLco). In any case, the method used must be in compliance with the European Respiratory Society (ERS)/American Thoracic Society(ATS) guideline on DLco measurements, and the prediction formula appropriate for that method.
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 7 | 8
Participants
  Change from baseline at week 12: Decrease by >10% | 2 | 1
  Change from baseline at week 12: Within 10% change | 5 | 7
  Change from baseline at week 12: Increase by >10% | 0 | 0
  Change from baseline at week 24: number analyzed (Participants) | 5 | 3
  Change from baseline at week 24: Decrease by >10% | 0 | 0
  Change from baseline at week 24: Within 10% change | 4 | 3
  Change from baseline at week 24: Increase by >10% | 1 | 0

12. Secondary Outcome: Change From Baseline in Daily Accelerometer Activity From Baseline at 12 and 24 Weeks: Score of Average Steps/Day
Description: Change from baseline in daily accelerometer activity from baseline at 12 and 24 weeks: Score of average Steps/day. Categories were defined as follows:
  Steps (total daily value) 0 = 0 to 1900 steps/day
  1. = 1901 to 3700 steps/day
  2. = 3701 to 5500 steps/day
  3. = 5501 to 7300 steps/day
  4. = >7301 steps/day
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 5 | 6
Score on a scale
  Change from baseline at week 12 | 0.4 (0.9) | 0.5 (0.5)
  Change from baseline at week 24: number analyzed (Participants) | 4 | 2
  Change from baseline at week 24 | -0.8 (1.7) | 0.0 (0.0)

13. Secondary Outcome: Change From Baseline in Daily Accelerometer Activity From Baseline at 12 and 24 Weeks: Score of Average Vector Magnitude Units (VMU)/Day
Description: Change from baseline in daily accelerometer activity from baseline at 12 and 24 weeks: Score of average vector magnitude units (VMU)/day. Categories were defined as follows:
  VMU (daily VMU/min) 0 = 0 to 50 VMU/min
  1. = 51 to 110 VMU/min
  2. = 111 to 190 VMU/min
  3. = 191 to 270 VMU/min
  4. = 271 to 440 VMU/min
  5. = >441 VMU/min
Time Frame: Baseline (day 1), week 12 (day 85) and week 24 (day 169).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
Number analyzed (Participants) | 5 | 6
Score on a scale
  Change from baseline at week 12 | 0.4 (0.9) | 0.3 (0.8)
  Change from baseline at week 24: number analyzed (Participants) | 4 | 2
  Change from baseline at week 24 | -0.5 (1.7) | -0.5 (0.7)

ADVERSE EVENTS:
Time Frame: From first Nintedanib drug intake on/after randomization (or re-start of nintedanib if interruption) to the last Nintedanib drug intake plus 28 days plus one day. Up to 263 days.
Description: Randomized set (RS): This patient set includes all randomized patients, whether treated with pulmonary rehabilitation or not.
Arm/Group | Nintedanib 150 mg | Nintedanib 150 mg + Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/9 | 1/10
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/10
Other Adverse Events (participants affected / at risk) | 4/9 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 mg (N=9) | Nintedanib 150 mg + Pulmonary Rehabilitation (N=10)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150 mg (N=9) | Nintedanib 150 mg + Pulmonary Rehabilitation (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lymphocyte percentage decreased (Investigations) | 0 | 1
Mean platelet volume decreased (Investigations) | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Trial was terminated prematurely due to difficulties with recruitment and a global BI recruitment hold implemented on 17 March 2020 because of the COVID-19 pandemic. The recruitment rate was slow and the target number of participants to be recruited was not reached. No inferential statistical analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT03717012/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT03717012/SAP_001.pdf